CLINICAL TRIAL: NCT05556057
Title: Feasibility of Mindfulness Meditation Training and Home Practice in Persons With Spinal Cord Injury: A Pilot Study
Brief Title: Feasibility of Mindfulness Meditation Training and Home Practice in Persons With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Sam Houston State University (Other); TIRR Memorial Hermann (Other)
Responsible Party: Principal Investigator, Radha Korupolu, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HSC-MS-22-0035; 1R34AT011530-01A1 (NIH)
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mindfulness meditation(MM) (Experimental)
  Interventions: Other: mindfulness meditation(MM)
- Health Education (Active Comparator)
  Interventions: Other: Health Education (active control)

INTERVENTIONS:
Other: mindfulness meditation(MM) — Participants will be provided with a unique invitation code that will allow them to download and use the free research version of the Mindfulness Coach app that is designed to deliver mindfulness training developed by the Veteran Affairs' National Center for PTSD.The app is tailored to users who may be skeptical about meditation practices by providing simple instructions and brief meditation exercises. The app offers written information about mindfulness as well as 12 audio-guided meditations each lasting 8-13 minutes, with an average length of 10 minutes
  Arms: mindfulness meditation(MM)
Other: Health Education (active control) — Participants will be asked to download and use the free TED Talk app.Each participant's account will include a list of over 80 TED Talks related to the six broad categories of sleep, nutrition, mood, relationships, chronic pain, and health behaviors. These talks range from 4 to 18 minutes and were reviewed/selected by the investigator team. The research coordinator(RC) will instruct them to watch or listen to these videos for ≥ 10 minutes daily for 6 days per week. The RC will ask participants to complete weekly logs of their TED Talk app use
  Arms: Health Education

SUMMARY:
The purpose of this study is to evaluate the feasibility and acceptability of a 6-week app-guided Mindfulness meditation training (MM) intervention and health education (active control) condition in people with spinal cord injury (SCI) who have chronic pain and to examine the feasibility of data collection procedures

DETAILED DESCRIPTION:
Our multidisciplinary, interinstitutional team of investigators proposes to randomize 60 SCI patients experiencing chronic pain to practice audio-guided MM for ≥ 10 minutes daily for 6 weeks using the free app "Mindfulness Coach" developed by the Department of Veteran Affairs, or to listen or view health education presentations (active control) ≥ 10 minutes daily for 6 weeks on the free TED app (active control). Primary outcomes are the feasibility and acceptability of proposed interventions in people with SCI and chronic pain. Secondary outcomes include the feasibility of collecting patient-reported outcomes of pain, anxiety, depression, mindfulness, quality of life, stress, fatigue and sleep disturbance.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic SCI of at least 6 months duration
* Chronic pain [defined as pain lasting at least 3 months with a pain intensity rating of 4 or higher on a 10-point visual analog scale]
* Understand spoken and written English sufficiently to provide informed consent
* participate in the intervention and complete study surveys

Exclusion Criteria:

* Lack of daily access to the internet using a smart phone or smart tablet
* Cognitive impairment (determined by their inability to demonstrate comprehension of informed consent by correctly answering 4 out of 5 questions pertaining to the study)
* Significant visual/hearing impairment that does not allow use of the MM app's audiovisual presentations or health education presentations on Ted-talk
* Use of any kind of meditation more than once a week in the last 3 months
* Inability to provide or obtain an email address for communication with study staff
* Inability to operate the app download or study related survey using a smartphone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Radha Korupolu, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Chelsea Ratcliff, PhD, Principal Investigator — Sam Houston State University
Locations (2):
- United States (2):
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - TIRR Memorial Hermann, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ratcliff CG, Lohiya S, Robinson-Whelen S, Taylor H, Ahn A, Korupolu R. Mindfulness buffers the association of pain with depression and anxiety among people with spinal cord injury: A cross-sectional study. Rehabil Psychol. 2024 Nov 11:10.1037/rep0000593. doi: 10.1037/rep0000593. Online ahead of print. PMID 39531687

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 70 participants screened 65 were eligible and enrolled. Of the 65 participants enrolled, 60 were randomized. 4 participants were unreachable prior to randomization and 1 participant withdrew before randomization.
Period: Overall Study
Arm/Group | Mindfulness Meditation(MM) | Health Education
Started | 29 | 31
Completed | 24 | 25
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Includes all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Meditation(MM) | Health Education | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.38 (14.97) | 47.65 (12.83) | 47.03 (13.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 20 | 21 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 27 | 26 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 19 | 21 | 40
  More than One Race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
  Do not wish to say | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 60
Education [Count of Participants; unit: Participants]
  Less than 12th grade | 1 | 2 | 3
  High School Graduate/ GED | 6 | 6 | 12
  Technical/Vocational school | 3 | 4 | 7
  Some College | 9 | 8 | 17
  Undergraduate Degree (BA/BS) | 9 | 4 | 13
  Graduate Degree (MA/Ph.D) | 1 | 7 | 8
Employment Status [Count of Participants; unit: Participants]
  Full time | 2 | 5 | 7
  Part-time | 1 | 3 | 4
  Retired | 8 | 8 | 16
  Unemployed | 18 | 15 | 33
Income [Count of Participants; unit: Participants]
  Under $15,000 | 6 | 1 | 7
  $15,000 to $24,999 | 6 | 3 | 9
  $25,000 to $34,999 | 5 | 1 | 6
  $35,000 to $49,999 | 3 | 3 | 6
  $50,000 to $74,999 | 1 | 7 | 8
  $75,000 to $99,999 | 2 | 4 | 6
  $100,000 & over | 2 | 2 | 4
  I do not wish to say | 0 | 4 | 4
  I do not know | 4 | 6 | 10
Marital status [Count of Participants; unit: Participants] — Population: Data for Marital status was not collected from 1 participant in the Health Education arm because they did not answer the question.
  Participants
    number analyzed (Participants) | 29 | 30 | 59
    Married | 7 | 9 | 16
    Widowed | 2 | 1 | 3
    Divorce or Separated | 6 | 9 | 15
    Living with significant other or partner | 5 | 1 | 6
    Single | 9 | 10 | 19
Cause of Spinal Cord Injury (Etiology) [Count of Participants; unit: Participants]
  Motor Vehicle Collision (MVC) | 14 | 14 | 28
  Falls | 1 | 6 | 7
  Sports | 2 | 3 | 5
  Assault | 7 | 6 | 13
  Medical/Surgical | 5 | 2 | 7
  Other Injury | 0 | 0 | 0
Mobility Status [Count of Participants; unit: Participants]
  Walk without assistance or an assistive device | 3 | 0 | 3
  Walk with assistance or assistive device (e.g., cane, walker, or braces) | 4 | 4 | 8
  Use manual/ hybrid wheelchair | 12 | 16 | 28
  Use a power wheelchair | 10 | 10 | 20
  Other | 0 | 1 | 1
Pain duration [Mean (Standard Deviation); unit: Months] | 7.39 (9.39) | 7.49 (6.37) | 7.44 (7.97)
Pain Type [Count of Participants; unit: Participants]
  Neuropathic pain | 21 | 23 | 44
  Nociceptive pain | 8 | 8 | 16
Neurological level [Count of Participants; unit: Participants] — The neurological level of injury is defined as the lowest segment of the spinal cord with normal sensory and motor function on both sides, based on the American Spinal Injury Association (ASIA) criteria. This level is determined by assessing key sensory points and motor functions. For this outcome, neurological levels are categorized as follows:
  Cervical (C1-C4)
  Cervical (C5-C8)
  Thoracic (T1-T5)
  Thoracic (T6-T12)
  Lumbar (L1-L5)
  Sacral
  Participants
    Cervical (C1-C4) | 5 | 3 | 8
    Cervical (C5-C8) | 14 | 12 | 26
    Thoracic (T1-T5) | 2 | 6 | 8
    Thoracic (T6-T12) | 5 | 7 | 12
    Lumbar (L1-L5) | 3 | 3 | 6
    Sacral | 0 | 0 | 0
Impairment [Count of Participants; unit: Participants] — Impairment is classified as either Complete or Incomplete based on the ASIA Impairment Scale (AIS).
  Complete impairment corresponds to AIS A, indicating a complete injury with no sensory or motor function is preserved in the sacral segments (S4-S5).
  Incomplete impairment corresponds to AIS B-D, where some sensory and/or motor function is preserved below the neurological level, including the sacral segments.
  Participants
    Complete | 7 | 14 | 21
    Incomplete | 20 | 17 | 37
    Unknown | 2 | 0 | 2
Pain intensity as assessed by the Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: score on a scale] — VAS pain scale is a range of scores from 0-10. A higher score indicates greater pain intensity.
  score on a scale | 6.69 (1.51) | 6.06 (1.50) | 6.36 (1.50)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Assessed by the Proportion of Eligible People Who Provide Consent
Time Frame: end of study at 3 years
Population: Overall Number of Participants Analyzed represents number of participants screened for study interest prior to enrollment.
Measure: Count of Participants; unit: Participants
Groups:
- All Eligible Participants: All eligible participants
Arm/Group | All Eligible Participants
Number analyzed (Participants) | 70
Participants | 65

2. Primary Outcome: Feasibility as Assessed by the Number of Participants Who Complete the Minimum Recommended Minutes (i.e., 60 Minutes/Per Week) of Using the MM or HE App During the 6 Weeks Intervention
Time Frame: post-intervention (6 weeks post-enrollment)
Population: Data were not collected from 5 participants in the Health Education arm because the 3 participants withdrew from the study and 2 participants were lost to follow up. Data were not collected from 5 participants in the mindfulness meditation arm because 4 participants were lost to follow up and 1 withdrew from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Meditation(MM) | Health Education
Number analyzed (Participants) | 24 | 26
Participants | 15 | 16

3. Primary Outcome: Feasibility as Assessed by the Number of Participants That Complete All Visits
Description: Number of participants that complete all visits defined as participants who completed all study assessments, including baseline visits, immediate post-intervention assessments, and 12-week follow-up assessments.
Time Frame: end of study (12 weeks post enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Meditation(MM) | Health Education
Number analyzed (Participants) | 24 | 25
Participants | 22 | 20

4. Primary Outcome: Acceptability Rate as Assessed by the Number of Participants Who Scored 20 or Greater on the Modified Client Satisfaction Questionnaire-8
Description: The Client Satisfaction Questionnaire-8 measures satisfaction and the total score ranges from 8 to 32. The greater the score the higher satisfaction.
Time Frame: post-intervention (6 weeks post-enrollment)
Population: Data were only collected from participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Meditation(MM) | Health Education
Number analyzed (Participants) | 22 | 19
Participants | 18 | 19

5. Primary Outcome: Feasibility as Assessed by the Number of Participants That Complete All Visits
Description: Number of participants that complete all visits defined as participants who completed all study assessments, including baseline visits and immediate post-intervention assessments.
Time Frame: post-intervention (6 weeks post-enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Meditation(MM) | Health Education
Number analyzed (Participants) | 24 | 25
Participants | 18 | 19

6. Secondary Outcome: Feasibility of Collecting Patient Reported Outcomes of Pain as Assessed by the Number of Participants Who Completed the International SCI Pain Basic Data Subset (Version 2)
Description: This survey contains 11 questions and each one is measured from 0(no pain) to 10(chronic pain),with a maximum score of 110, a higher number indicating more pain
Time Frame: Baseline
Population: Feasibility outcome measures were pre-specified to be collected as a single group at baseline, this data was collected prior to randomization. Enrolled participants are defined as those who provided informed consent prior to randomization.
Measure: Count of Participants; unit: Participants
Groups:
- All Enrolled Participants: All enrolled participants are those who provided informed consent
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 65
Participants | 60

7. Secondary Outcome: Feasibility of Collecting Patient Reported Outcomes of Pain as Assessed by the Number of Participants Who Completed the International SCI Pain Basic Data Subset (Version 2)
Description: as for outcome 6
Time Frame: post-intervention (6 weeks post-enrollment), end of study (12 weeks post enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Meditation(MM) | Health Education
Number analyzed (Participants) | 24 | 25
Participants
  post-intervention (6 weeks post-enrollment) | 18 | 19
  end of study (12 weeks post enrollment) | 22 | 20

8. Secondary Outcome: Feasibility of Collecting Patient Reported Outcomes of Pain-related Distress as Assessed by the Number of Participants Who Completed the Chronic Pain Acceptance Questionnaire (CPAQ-R8)
Description: This is a 20 item questionnaire, each is scored from 0(never true) to 6(always true), a higher number indicating higher acceptance
Time Frame: baseline
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 65
Participants | 60

9. Secondary Outcome: Feasibility of Collecting Patient Reported Outcomes of Pain-related Distress as Assessed by the Number of Participants Who Completed the Chronic Pain Acceptance Questionnaire (CPAQ-R8)
Description: as for outcome 8
Time Frame: post-intervention (6 weeks post-enrollment), end of study (12 weeks post enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Meditation(MM) | Health Education
Number analyzed (Participants) | 24 | 25
Participants
  post-intervention (6 weeks post-enrollment) | 20 | 19
  end of study (12 weeks post enrollment) | 23 | 22

10. Secondary Outcome: Feasibility of Collecting Patient Reported Outcomes of Brief Pain as Assessed by the Number of Participants Who Completed the Brief Pain Catastrophizing Scale (Brief PCS)
Description: This measures three aspects of catastrophic cognitions about pain-rumination, magnification, and helplessness. This is a 13 item questionnaire. Each question has five response options ranging from 0 (not at all) to 4 (all the time) scale, with a maximum score of 52
Time Frame: Baseline
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 65
Participants | 60

11. Secondary Outcome: Feasibility of Collecting Patient Reported Outcomes of Brief Pain as Assessed by the Number of Participants Who Completed the Brief Pain Catastrophizing Scale (Brief PCS)
Description: as for outcome 10
Time Frame: post-intervention (6 weeks post-enrollment), end of study (12 weeks post enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Meditation(MM) | Health Education
Number analyzed (Participants) | 24 | 25
Participants
  post-intervention (6 weeks post-enrollment) | 20 | 19
  end of study (12 weeks post enrollment) | 23 | 22

12. Secondary Outcome: Feasibility of Collecting Patient Reported Outcomes of Anxiety as Assessed by the Number of Participants Who Completed the General Anxiety Disorder-7 (GAD-7) Questionnaire
Description: This is an 7 item questionnaire, each is scored from 0(not at all) to 3(nearly every day), a higher score indicating more anxiety
Time Frame: Baseline
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 65
Participants | 64

13. Secondary Outcome: Feasibility of Collecting Patient Reported Outcomes of Anxiety as Assessed by the Number of Participants Who Completed the General Anxiety Disorder-7 (GAD-7) Questionnaire
Description: as for outcome 12
Time Frame: post-intervention (6 weeks post-enrollment), end of study (12 weeks post enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Meditation(MM) | Health Education
Number analyzed (Participants) | 24 | 25
Participants
  post-intervention (6 weeks post-enrollment) | 20 | 19
  end of study (12 weeks post enrollment) | 23 | 22

14. Secondary Outcome: Feasibility of Collecting Patient Reported Outcomes of Depression as Assessed by the Number of Participants Who Completed the Patient Health Questionnaire (PHQ-8)
Description: This is an 8 item questionnaire.Each question is scored from 0 to 1 day = "not at all," 2 to 6 days = "several days," 7 to 11 days = "more than half the days," and 12 to 14 days = "nearly every day". Total score is determined by adding together the scores of each of the four items. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12).
Time Frame: Baseline
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 65
Participants | 64

15. Secondary Outcome: Feasibility of Collecting Patient Reported Outcomes of Depression as Assessed by the Number of Participants Who Completed the Patient Health Questionnaire (PHQ-8)
Description: as for outcome 14
Time Frame: post-intervention (6 weeks post-enrollment), end of study (12 weeks post enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Meditation(MM) | Health Education
Number analyzed (Participants) | 24 | 25
Participants
  post-intervention (6 weeks post-enrollment) | 20 | 19
  end of study (12 weeks post enrollment) | 23 | 22

16. Secondary Outcome: Feasibility of Collecting Patient Reported Outcomes of Mindfulness as Assessed by the Number of Participants Who Completed the Five Facet Mindfulness Questionnaire-15 (FFMQ-15)
Description: This is a 15 item questionnaire, each is scored from 1(never or very rarely true) to 5(very often or always true) for a maximum score of 120, higher score indicating more mindfulness
Time Frame: Baseline
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 65
Participants | 64

17. Secondary Outcome: Feasibility of Collecting Patient Reported Outcomes of Mindfulness as Assessed by the Number of Participants Who Completed the Five Facet Mindfulness Questionnaire-15 (FFMQ-15)
Description: as for outcome 16
Time Frame: post-intervention (6 weeks post-enrollment), end of study (12 weeks post enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Meditation(MM) | Health Education
Number analyzed (Participants) | 24 | 25
Participants
  post-intervention (6 weeks post-enrollment) | 20 | 19
  end of study (12 weeks post enrollment) | 23 | 22

18. Secondary Outcome: Feasibility of Collecting Patient Reported Outcomes of Quality of Life as Assessed by the Number of Participants Who Completed the SCI-quality of Life (QOL): Positive Affect and Well Being-Short Form (PAWB-SF)
Description: This is a 10 item scale each scored from (1)never to (5)always, with a maximum score of 50 a higher number indicating a better outcome
Time Frame: Baseline
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 65
Participants | 64

19. Secondary Outcome: Feasibility of Collecting Patient Reported Outcomes of Quality of Life as Assessed by the Number of Participants Who Completed the SCI-quality of Life (QOL): Positive Affect and Well Being-Short Form (PAWB-SF)
Description: as for outcome 18
Time Frame: post-intervention (6 weeks post-enrollment), end of study (12 weeks post enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Meditation(MM) | Health Education
Number analyzed (Participants) | 24 | 25
Participants
  post-intervention (6 weeks post-enrollment) | 20 | 19
  end of study (12 weeks post enrollment) | 23 | 22

20. Secondary Outcome: Feasibility of Collecting Perceived Stress as Assessed by the Number of Participants Who Completed the Perceived Stress Scale (PSS-4)
Description: The Perceived Stress Scale (PSS-4) is a four-item scale, each item is scored from 0(never) to 4(very often). The total score ranges from 0 to 16, a higher score indicating more stress
Time Frame: Baseline
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 65
Participants | 64

21. Secondary Outcome: Feasibility of Collecting Perceived Stress as Assessed by the Number of Participants Who Completed the Perceived Stress Scale (PSS-4)
Description: as for outcome 20
Time Frame: post-intervention (6 weeks post-enrollment), end of study (12 weeks post enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Meditation(MM) | Health Education
Number analyzed (Participants) | 24 | 25
Participants
  post-intervention (6 weeks post-enrollment) | 20 | 19
  end of study (12 weeks post enrollment) | 23 | 22

22. Secondary Outcome: Feasibility of Collecting Fatigue as Assessed by the Number of Participants Who Completed the PROMIS Fatigue- Short Form 4a
Description: Each question has five response options ranging in value from five (very poor) to one (very good), a higher number indicating more fatigue.
Time Frame: Baseline
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 65
Participants | 64

23. Secondary Outcome: Feasibility of Collecting Fatigue as Assessed by the Number of Participants Who Completed the PROMIS Fatigue- Short Form 4a
Description: as for outcome 22
Time Frame: post-intervention (6 weeks post-enrollment), end of study (12 weeks post enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Meditation(MM) | Health Education
Number analyzed (Participants) | 24 | 25
Participants
  post-intervention (6 weeks post-enrollment) | 20 | 19
  end of study (12 weeks post enrollment) | 23 | 22

24. Secondary Outcome: Feasibility of Collecting Psychological Inflexibility/Experiential Avoidance as Assessed by the Number of Participants Who Completed the Acceptance and Action Questionnaire (AAQ-2)
Description: This contains 7 items and answers are given on a 7-point scale ranging from 1 (never true) to 7 (always true). High scores on the AAQ-2 are reflective of greater experiential avoidance and immobility, while low scores reflect greater acceptance and action.
Time Frame: Baseline
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 65
Participants | 64

25. Secondary Outcome: Feasibility of Collecting Psychological Inflexibility/Experiential Avoidance as Assessed by the Number of Participants Who Completed the Acceptance and Action Questionnaire (AAQ-2)
Description: as for outcome 24
Time Frame: post-intervention (6 weeks post-enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Meditation(MM) | Health Education
Number analyzed (Participants) | 24 | 25
Participants | 20 | 19

26. Secondary Outcome: Feasibility of Collecting Psychological Inflexibility/Experiential Avoidance as Assessed by the Number of Participants Who Completed the Acceptance and Action Questionnaire (AAQ-2)
Description: as for outcome 24
Time Frame: end of study (12 weeks post enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Meditation(MM) | Health Education
Number analyzed (Participants) | 24 | 25
Participants | 23 | 22

27. Secondary Outcome: Feasibility of Collecting Sleep Disturbance as Assessed by the Number of Participants Who Completed the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance- Short Form 4a
Description: This is a 4 item questionnaire and each question has five response options ranging in value from five (very poor) to one (very good) for a maximum score of 16, higher number indicating worse outcome.
Time Frame: Baseline
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 65
Participants | 64

28. Secondary Outcome: Feasibility of Collecting Sleep Disturbance as Assessed by the Number of Participants Who Completed the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance- Short Form 4a
Description: as for outcome 27
Time Frame: post-intervention (6 weeks post-enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Meditation(MM) | Health Education
Number analyzed (Participants) | 24 | 25
Participants | 20 | 19

29. Secondary Outcome: Feasibility of Collecting Sleep Disturbance as Assessed by the Number of Participants Who Completed the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance- Short Form 4a
Description: as for outcome 27
Time Frame: end of study (12 weeks post enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Meditation(MM) | Health Education
Number analyzed (Participants) | 24 | 25
Participants | 23 | 22

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Mindfulness Meditation(MM) | Health Education
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 2/29 | 1/31
Other Adverse Events (participants affected / at risk) | 1/29 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mindfulness Meditation(MM) (N=29) | Health Education (N=31)
Hospitalized due to spinal cord injury complications (Nervous system disorders) | 2 | 0
Surgery (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mindfulness Meditation(MM) (N=29) | Health Education (N=31)
Urinary tract infection (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT05556057/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT05556057/ICF_001.pdf